CLINICAL TRIAL: NCT02203461
Title: Changes in Insulin Resistance in Healthy Volunteers on STRIBILD® Medication - A Controlled, Mono Center, Three-arm, Randomized Phase I Study.
Brief Title: Changes in Insulin Resistance in Healthy Volunteers on STRIBILD® Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Gilead Sciences (Industry); MUC Research GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR-1383--0030-I; 2014-000359-98 (EudraCT Number)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Insulin Resistance
Keywords: ART, HIV, insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Lopinavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Experimental): STRIBILD® Tenofovir disaproxil fumarate/emtricitabine/elvitegravir/cobicistat
  Interventions: Drug: Tenofovir disaproxil fumarate/emtricitabine/elvitegravir/cobicistat
- Group II (Active Comparator): Truvada®/Kaletra® Tenofovir disaproxil fumarate/emtricitabine + Lopinavir/ritonavir
  Interventions: Drug: Tenofovir disaproxil fumarate/emtricitabine + Lopinavir/ritonavir
- Group III (Experimental): Truvada®/Prezista®/Norvir® Tenofovir disaproxil fumarate/emtricitabine + ritonavir-boosted darunavir
  Interventions: Drug: Tenofovir disaproxil fumarate/emtricitabine + ritonavir-boosted darunavir

INTERVENTIONS:
Drug: Tenofovir disaproxil fumarate/emtricitabine/elvitegravir/cobicistat — STRIBILD® QD, d1-14
  Other Names: STRIBILD®
  Arms: Group I
Drug: Tenofovir disaproxil fumarate/emtricitabine + Lopinavir/ritonavir — Truvada®/ Kaletra® 200/50 mg QD, d1-14
  Other Names: Truvada® / Kaletra®
  Arms: Group II
Drug: Tenofovir disaproxil fumarate/emtricitabine + ritonavir-boosted darunavir — Truvada®/Prezista® 800 mg/Norvir®100 mg Medication, QD, d1-14
  Other Names: Truvada®/Prezista®/Norvir®
  Arms: Group III

SUMMARY:
Changes in insulin resistance in healthy volunteers with normal body weight (BMI 18-25) after 14 days of STRIBILD®-, Truvada®/Kaletra® or Truvada®/Prezista®/Norvir® intake, measured by hyperinsulinemic euglycemic clamp.

DETAILED DESCRIPTION:
The measurement of insulin resistance will be performed in 30 HIV-negative healthy non-obese (BMI 18-25) male volunteers before and after 14 days (+/- 2 days) of treatment with STRIBILD® (treatment 1, n=10), as compared to TVD, LPV/r (treatment 2, n=10) and TVD, DRV/r (treatment 3, n=10). The volunteers will be randomly assigned to one of three groups. The measurement of insulin resistance, lipid and glucose metabolism will be performed; before and immediately after the treatment. Furthermore, the therapy compliance will be verified using the method of drug counting and therapeutic drug monitoring (TDM).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age 18-40 years
* Informed consent and willingness in study participation
* Birth control during study period

Exclusion Criteria:

* Participation in other clinical trials
* Contraindication or known allergy to study medication
* Known metabolic disease incl. Diabetes mellitus, Hypertriglyceridemia or others
* Known alcohol or nicotine abuse
* HIV infection
* History of pharmaceutical study in the last 4 weeks
* BMI < 18 > 25
* Long-term or regular medication
* Known liver-, renal-, cardiovascular, lung, gastrointestinal, endocrine, neurologic, psychiatric or metabolic disorder
* Dependence to study center or coordinator
* Inmates or psychiatric treatment

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in insulin resistance, measured by hyperinsulinemic euglycemic clamp | Day 14
  Changes in insulin resistance in healthy volunteers with normal body weight (BMI 18-25) after 14 days of STRIBILD®-, Truvada®/Kaletra® or Truvada®/Prezista®/Norvir® intake, measured by hyperinsulinemic euglycemic clamp.

SECONDARY OUTCOMES:
Changes in metabolic parameters | Day 14
  Changes in lipid, metabolic hormons and "HOMA-IR", "Homa-beta", "QUICKIE" test.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph D Spinner, MD, Principal Investigator — University Hospital Klinikum rechts der Isar, Technische Universitaet Muenchen
Locations (1):
- University Hospital Klinikum rechts der Isar (TUM), Munich, Bavaria, Germany